CLINICAL TRIAL: NCT03185039
Title: Study of the Predictive Impact of MMP2 and MMP9 Levels for Patients With Metastatic Kidney Cancer Treated With Anti-angiogenic Agents Compared to Patients Not Treated With Antiangiogenic (Localized Kidney Cancer and Oligometastatic)
Brief Title: Predictive Impact of MMP2 and MMP9 Levels for Patients With Metastatic Kidney Cancer Treated With Anti-angiogenic Agents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MMP-Rein-IPC 2015-029
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- kidney cancer (Experimental): Localized, oligometastatic or metastatic
  Interventions: Procedure: Blood and tumor samples

INTERVENTIONS:
Procedure: Blood and tumor samples — Blood and tumor samples

SUMMARY:
Prospective research of Matrix Metalloproteinases (MMP) 2 and 9 as predictive biomarkers in metastatic kidney cancer patients treated with 2 anti angiogenic agents (Sunitinib or Pazopanib).

DETAILED DESCRIPTION:
The objective is to analyze the predictive impact of circulating MMP2 and MMP9 on the progression-free survival of patients with metastatic kidney cancer treated with anti-angiogenic agents (Sunitinib or Pazopanib) in comparison with two untreated cohorts (localized or oligometastatic cancer).

Prospective monocenter, open-label study

In the frame of disease management blood samples will be collected at different times of follow-up regarding disease status (localized, oligometastatic and metastatic) and tissue samples will be collected for patients scheduled for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient male or female, aged of more than 18 years
2. Patient with any of the following conditions:

   * Kidney cancer localized at diagnosis.
   * Metastatic kidney cancer when anti-angiogenic therapy is initiated by Sunitinib or Pazopanib
   * Oligometastatic kidney cancer without systemic treatment (local treatment)
3. ECOG = 0 to 2
4. Patient affiliated to, or beneficiary of, the national social security.
5. Patient having signed informed consent

Exclusion Criteria:

1. Patient previously treated with anti-angiogenic agents.
2. Person in an emergency situation, adult subject to a legal protection measure (a guardian, guardianship or safeguard of justice), or unable of expressing his / her consent.
3. Impossibility to undergo the medical follow-up of the trial for geographical, social or psychological reasons 4. History of malignant disease in the 5 years prior to inclusion (except basal cell carcinoma of the skin or epithelioma of the cervix in situ, or prostate cancer with a good prognosis (stage T <3 and Gleason <7)) accidentally discovered during the histological analysis of the tumor sample.

5- Pregnant or nursing women 6- Contraindications to the procedure of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05-29 (Actual); Primary Completion 2022-12-13 (Estimated); Study Completion 2022-12-13 (Estimated)

PRIMARY OUTCOMES:
Plasma level of the MMP2 and MMP9 markers | at initial sampling
  ELISA assay
Survival without progression | Up to 18 months
  date of progression (RECIST criteria), date of death

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jubb AM, Harris AL. Biomarkers to predict the clinical efficacy of bevacizumab in cancer. Lancet Oncol. 2010 Dec;11(12):1172-83. doi: 10.1016/S1470-2045(10)70232-1. PMID 21126687
- [Result] Tabouret E, Boudouresque F, Barrie M, Matta M, Boucard C, Loundou A, Carpentier A, Sanson M, Metellus P, Figarella-Branger D, Ouafik L, Chinot O. Association of matrix metalloproteinase 2 plasma level with response and survival in patients treated with bevacizumab for recurrent high-grade glioma. Neuro Oncol. 2014 Mar;16(3):392-9. doi: 10.1093/neuonc/not226. Epub 2013 Dec 9. PMID 24327581
- [Result] Tabouret E, Boudouresque F, Farina P, Barrie M, Bequet C, Sanson M, Chinot O. MMP2 and MMP9 as candidate biomarkers to monitor bevacizumab therapy in high-grade glioma. Neuro Oncol. 2015 Aug;17(8):1174-6. doi: 10.1093/neuonc/nov094. No abstract available. PMID 26142442
- [Result] Tabouret E, Bertucci F, Pierga JY, Petit T, Levy C, Ferrero JM, Campone M, Gligorov J, Lerebours F, Roche H, Bachelot T, van Laere S, Ueno NT, Toiron Y, Finetti P, Birnbaum D, Borg JP, Viens P, Chinot O, Goncalves A. MMP2 and MMP9 serum levels are associated with favorable outcome in patients with inflammatory breast cancer treated with bevacizumab-based neoadjuvant chemotherapy in the BEVERLY-2 study. Oncotarget. 2016 Apr 5;7(14):18531-40. doi: 10.18632/oncotarget.7612. PMID 26921265
- See also: Official website of the sponsor — http://institutpaolicalmettes.fr